CLINICAL TRIAL: NCT03185975
Title: Providing Online Counseling for Home-Based HIV Testing With Transgender Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Robert Stephenson, Professor, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HUM00123412
Record Dates: First submitted 2017-06-11; First posted 2017-06-14 (Actual); Last update posted 2019-10-21 (Actual); Status verified 2019-10

CONDITIONS: Hiv; Transgender Youth
Keywords: HIV; transgender; trans; youth; home testing
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Motivational Interviewing; Referral and Consultation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Placebo Comparator): Each participant will receive an at-home test kit and will be asked to test and return results to investigator.
  Interventions: Behavioral: at-home test kit
- Intervention Arm (Active Comparator): Each participant will receive an at-home test kit and will be asked to take the test in conjunction with an online Motivational interviewing/certified testing and referral (MI/CTR).
  Interventions: Behavioral: Motivational Interviewing and Certified Testing and Referral

INTERVENTIONS:
Behavioral: at-home test kit — Transgender youth in the control arm will receive test kits, but will not receive any testing intervention. Once individual results are reported, participants will be contacted via phone or email by study staff with options for referrals to services. Participants will complete follow-up surveys at 3, 6, 9, and 12 months post-testing.
  Arms: Control arm
Behavioral: Motivational Interviewing and Certified Testing and Referral — Transgender individuals randomized to the experimental group (MI/CTR) will receive HIV counseling and testing via an online, HIPPA-compliant videoconferencing service. The session will last less than one hour and focus on HIV testing, prevention strategies, and/or linkage to HIV care, depending on the individual's test results. Participants will complete follow up surveys at 3, 6, 9 and 12 months.
  Other Names: MICTR MI/CTR
  Arms: Intervention Arm

SUMMARY:
This research study will recruit 200 transgender youths between the ages of 15-24. There are two arms to the research study: the control and the intervention arm. Each eligible participant will be randomized into either arm. The control arm participants receive an OraQuick HIV testing kit sent to an address of their choice and instructions of how to conduct the test. They will enter their results on the research study website and complete surveys at 3 month intervals until an entire year has passed. Participants in the intervention arm will receive an OraQuick HIV testing kit sent to them and will receive video-based counseling called Motivational Interviewing and Certified Testing and Referral. After this counseling session, the results from the OraQuick HIV test will be logged by study staff. Then, participants in the intervention arm will fill out surveys at 3 month intervals until a year has passed.

ELIGIBILITY:
Inclusion Criteria:

* male sex at birth, identifies as female, trans feminine, trans woman, female
* female sex at birth, identifies as male, trans male, trans masculine, male
* agender, genderfluid, genderqueer
* between the ages of 15-24,
* negative or unknown HIV status and not having tested in the least 3 months
* willingness to have HIV test kit delivered to an address they provide
* wilingness to be tested for HIV
* willingness to be randomized to either study arm
* willingness and ability to participate in video-based counseling (must have a computer or tablet with video and audio capabilities, internet access)

Exclusion Criteria:

* same sex assigned at birth and currently identifies as that same sex
* aged 14 years or younger, or 25 years or older
* reports having a positive HIV status during the baseline survey or screener survey before testing unwillingness to have HIV test kit delivered to an address they provide
* unwillingness to test for HIV
* unwillingness to be randomized
* unwillingness or inability to participate in video-based counseling

Ages: 15 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — must have a differing gender identity than what was reported as the sex assigned at birth, intersex, agender, genderqueer, and genderfluid individuals are also eligible regardless of their sex assigned at birth.
Enrollment: 200 (Actual)
Dates: Start 2017-06-19 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Increase uptake of HIV testing for transgender youth | 1 year
  Assess differences and changes in TY's sexual-risk behaviors between those who receive the home-testing with video-based MI/CTR (intervention arm) compared to those who receive the home-testing alone (control arm). 200 TY (100 male: 100 female) will be randomized to either the intervention or control arm and followed for 6 months with surveys taken at baselines and months 3, 6, 9 and 12 months.

SECONDARY OUTCOMES:
Changes in Sexual Behavior | 1 year.
  We measure changes in sexual behavior using behavioral measures based on information collected from the baseline survey, MI/CTR session for the intervention arm participants, and subsequent surveys each 3 months until one year from the initial survey has occurred.
Linkage to Care | 1 year
  We will measure linkage to care with the following outcomes as indicators per the recent recommendations of the Institute of Medicine and CDC: within 3 months of HIV diagnosis, attending at least one clinical care appointment, having at least one CD4 test performed and having at least one viral load test performed.

CONTACTS AND LOCATIONS:
Overall Officials: Rob Stephenson, PhD, Principal Investigator — University of Michigan Center for Sexuality & Health Disparities
Locations (1):
- University of Michigan Center for Sexuality and Health Disparities, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Stephenson R, Todd K, Kahle E, Sullivan SP, Miller-Perusse M, Sharma A, Horvath KJ. Project Moxie: Results of a Feasibility Study of a Telehealth Intervention to Increase HIV Testing Among Binary and Nonbinary Transgender Youth. AIDS Behav. 2020 May;24(5):1517-1530. doi: 10.1007/s10461-019-02741-z. PMID 31760536
- [Derived] Stephenson R, Metheny N, Sharma A, Sullivan S, Riley E. Providing Home-Based HIV Testing and Counseling for Transgender Youth (Project Moxie): Protocol for a Pilot Randomized Controlled Trial. JMIR Res Protoc. 2017 Nov 28;6(11):e237. doi: 10.2196/resprot.8562. PMID 29183868